CLINICAL TRIAL: NCT03510130
Title: Routine Maternal Leg Movements During the Second Stage and the Rate of Operative Deliveries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0553-17-RMB
Record Dates: First submitted 2018-03-11; First posted 2018-04-27 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Cesarean Delivery Affecting Fetus or Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine leg movement (Experimental): Intervention group- In the second stage of labor, attending physician or nurse will help the participant in routine leg movements every 20-30 minutes.
  Interventions: Other: Routine leg movement
- Control group (No Intervention): Control group which includes women during the second stage of labor with no intervention (routine leg movement).

INTERVENTIONS:
Other: Routine leg movement — Routine leg movement to the right and left in the supine position during the second stage of labor, for 3 minutes every 20-30 minutes by the attending physician or nurse.
  Arms: Routine leg movement

SUMMARY:
Cesarean delivery rates have risen in the US in a dramatic fashion from less than 5% in the 1960 to 32.7% by 2013 with stable rate around 32-33% in the last five years , cesarean delivery is associated with increased maternal morbidity and mortality, Labor arrest is the most common indication for cesarean delivery, Maternal position during the second stage of labor has been suggested to affect the risk of instrumental vaginal delivery. A Cochrane review of position in the second stage of labor in women without epidural showed a reduction in instrumental vaginal delivery in the upright group, although the quality of the included trials was reported to be generally poor, A Cochrane review of position in the second stage of labour for women with epidural analgesia was published in 2017, This review included trials that compared upright with recumbent positions and suggested no effect.

No prior studies examined whether maternal legs movement during the second stage of labor has any effect on the rate of operative deliveries.

DETAILED DESCRIPTION:
A randomized controlled trial to determine whether routine maternal leg movement during the second stage of labor decreases the rate of operative deliveries (instrumental delivery of cesarean section )

ELIGIBILITY:
Inclusion Criteria:

•Women who had a low risk pregnancy followed by an uncomplicated vaginal delivery, instrumental delivery or cesarean section.

Exclusion Criteria:

•Women who had a high risk pregnancy ((IUGR, hypertension disorders of pregnancy, maternal cardiovascular or respiratory illness).

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Obstetrical study
Enrollment: 300 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Routine legs movement during the second stage of labor and the rates of cesarean deliveries (In percentage of the total deliveries) and instrumental deliveries (In percentage of total deliveries) | up to 12 months
  The study objective is to determine whether routine maternal leg movement during the second stage of labor decreases the rate of operative deliveries (instrumental and cesarean deliveries)

IPD SHARING:
Plan to Share IPD: No